CLINICAL TRIAL: NCT03728894
Title: Oral Sedation With/Without Nitrous Oxide in Pediatric Dental Patients
Brief Title: Oral Sedation With and Without Nitrous Oxide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Principal Investigator, Nabih Raslan, Principal investigator, Tishreen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Tishreen-sedation
Record Dates: First submitted 2018-10-26; First posted 2018-11-02 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Behavior, Child
Keywords: Midazolam; hydroxyzine; oxygen; behavior; child; tooth
MeSH Terms: conditions — Child Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: blinded, randomized controlled trial, comparing two groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor) Each of the children/parents, the dentist and the outcomes assessors were blinded. To ensure the blindness of the dentist, the inhalation sedation machine was placed in a way that he could not see the flow rate panel or the type of the administered gases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Midazolam-hydroxyzine with 100% O2 (Active Comparator): Midazolam-hydroxyzine with 100% O2 was administrated to 30 children. Drug: Oral Medication (midazolam 7.5 mg and hydroxyzine 10 mg) and Inhalation Gas 100% O2 Patients were randomly assigned to received one of two regimens (A,B) in across over design, Behavior was assessed using the modified Houpt behavioral rating scale, by evaluating the videotapes of all patients at both the pretreatment and treatment phases.
  Interventions: Drug: Midazolam-hydroxyzine with 100% O2
- Midazolam-hydroxyzine with 50% N2O/ O2 (Experimental): children received Midazolam-hydroxyzine with 50% N2O/O2, one tablet of oral midazolam 7.5 mg and one tablet of hydroxyzine 10 mg with 50% N2O/O2. Drug: Oral Medication and Inhalation Gas Patients were randomly assigned to received one of two regimens (A,B) in across over design, Behavior was assessed using the modified Houpt behavioral rating scale, by evaluating the videotapes of all patients at both the pretreatment and treatment phases.
  Interventions: Drug: Midazolam-hydroxyzine with 50% N2O/O2

INTERVENTIONS:
Drug: Midazolam-hydroxyzine with 100% O2 — Patients received Oral Sedatives with 100% O2 ,Behavior was assessed using the modified Houpt behavioral rating scale, by evaluating the videotapes of all patients at both the pretreatment and treatment phases.
  Other Names: A
  Arms: A: Midazolam-hydroxyzine with 100% O2
Drug: Midazolam-hydroxyzine with 50% N2O/O2 — Patients received Oral Sedatives with 50% nitrous ,Behavior was assessed using the modified Houpt behavioral rating scale, by evaluating the videotapes of all patients at both the pretreatment and treatment phases.
  Other Names: B
  Arms: Midazolam-hydroxyzine with 50% N2O/ O2

SUMMARY:
Aims: The objective of the current study was to evaluate the effectiveness of oral midazolam-hydroxyzine with/without nitrous oxide. Design: This was a randomized split mouth, cross over and triple-blinded clinical study. Thirty uncooperative healthy children aged six to nine, whose needed dental treatments.

DETAILED DESCRIPTION:
The purpose of this study was to compare the efficacy of combining oral midazolam-hydroxyzine with/without N2O/O2 in sedating uncooperative schoolchildren undergoing dental treatment. Thirty uncooperative healthy children aged six to nine were randomly selected to receive either one tablet of oral midazolam 7.5 mg and one tablet of hydroxyzine 10 mg with 100% O2 (regimen A), or one tablet of oral midazolam 7.5 mg and one tablet of hydroxyzine 10 mg with 50% N2O/O2 (regimen B) in a crossover design. Behavior was assessed using the modified Houpt behavioral rating scale, by evaluating the videotapes of all patients at both the pretreatment phase (injection, rubber dam RD, operating high-speed handpiece with touching the tooth without drilling) and the treatment phase (drilling, restoration).

ELIGIBILITY:
Criteria: Inclusion Criteria:

* ASA Classification I.
* minimum weight of 18 kg
* uncooperative children scored 1 or 2 on Frankle Scale.
* requiring nonemergency, bilateral mandibular dental treatments under local anesthesia.

Exclusion Criteria:

* known allergy to midazolam and/or hydroxyzine.
* upper respiratory tract infection with nasal discharge.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-01-06 (Actual); Study Completion 2019-01-06 (Actual)

PRIMARY OUTCOMES:
Behavior improvement on the modified Houpt behavioral rating scale | Behavior will assess at the end of the session (about 30-90 min) by evaluating the sessions 's videotapes using overall assessment (range from 1 to 4, higher values represent a better outcome) of the modified Houpt behavioral rating scale
  Behavior assessment improvement related to the addition of N2O/O2 to the combination midazolam-hydroxyzine.
Behavior improvement on the modified Houpt behavioral rating scale | Behavior assess after 30 min of oral medications administered by evaluate the sessions's videotapes using of Sleep,movement,Head/oral resistance,Cry,Verbal assessments(range1- 4,higher values is the better outcome)of modified Houpt behavioral scale
  Behavior assessment improvement related to the addition of N2O/O2 to the combination midazolam-hydroxyzine.

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Dr, Study Chair — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided
up to date, there is no decision about IPD sharing.